CLINICAL TRIAL: NCT05317689
Title: Comparison of the Effects of PEX20 (Oral Psilocin), PEX30 (Sublingual Psilocin), and PEX10 (Oral Psilocybin) in Healthy Adults
Brief Title: Comparing the Effects of Psilocin and Psilocybin in Healthy Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Filament Health Corp. (Industry)
Responsible Party: Principal Investigator, Joshua Woolley, MD, PhD, Associate Professor, Psychiatry, University of California, San Francisco
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: IRB#21-33765; PR#202143H (Other: Research Advisory Panel - California); 156917 (Other: FDA)
Record Dates: First submitted 2022-03-07; First posted 2022-04-08 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: Psilocybin; Psilocin; Psilocybin Therapy; Psychedelics; Healthy; San Francisco
MeSH Terms: interventions — psilocin; Psilocybin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral & Sublingual Psilocin, & Oral Psilocybin (Active Comparator): Every participant will be administered Oral Psilocin, Sublingual Psilocin, and oral psilocybin in a randomized order.
  Interventions: Drug: Psilocin; Drug: Psilocybin; Drug: Sublingual Psilocin
- Sublingual Psilocin (Active Comparator): Depending on a number of factors, participants may complete a fourth session where they receive sublingual psilocin for the second time.
  Interventions: Drug: Sublingual Psilocin

INTERVENTIONS:
Drug: Psilocin — 17.5mg oral psilocin with psychological support and physiological monitoring
  Arms: Oral & Sublingual Psilocin, & Oral Psilocybin
Drug: Psilocybin — 25mg oral psilocybin with psychological support and physiological monitoring
  Arms: Oral & Sublingual Psilocin, & Oral Psilocybin
Drug: Sublingual Psilocin — 2.18mg - 4.36mg sublingual psilocin with psychological support and physiological monitoring

SUMMARY:
To compare the physiological and psychological effects of psilocin taken orally by pill or sublingually by dissolving a tablet under the tongue to those of psilocybin taken by pill in healthy adults.

DETAILED DESCRIPTION:
The primary goal of this study is to compare the physiological and psychological effects of psilocin taken orally by pill or sublingually dissolved under the tongue to those of psilocybin taken by pill. Twenty participants, ages 25 to 50, with one previous experience with psychedelics, and who meet all other inclusion and exclusion criteria at screening will be enrolled. After baseline assessments, participants will engage in preparatory visits with trained facilitators, followed by drug administration, supervised by the facilitators and a clinician who will conduct safety monitoring throughout. Participants will then complete assessment and integration sessions with the facilitators in order to help process the experience. The same preparation, procedures, integration, and supervision will be repeated up to three more times with each participant.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 to 50
* Comfortable speaking and writing in English
* Commit to attending all study visits and remote data collection tasks
* No planned surgeries during the study
* Had at least one prior experience with a psychedelic substance
* Generally mentally and physically healthy
* Agree to abstain from THC, CBD, or nicotine products during study

Exclusion Criteria:

* Participated in another clinical trial within 30 days of entry to this trial
* Regular use of medications that may have problematic interactions with psilocybin, including but not limited to dopamine agonists, MAO inhibitors, N-methyl-D-aspartate (NMDAR) antagonists, antipsychotics, and stimulants
* A health condition that makes study unsafe or unfeasible, determined by study physicians

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Physiological Effects | Baseline to 8 hours following drug delivery
  blood pressure
Physiological Effects | Baseline to 8 hours following drug delivery
  heart rate
Psychological Effects | Baseline to 4 weeks after drug delivery
  - Peak psychedelic intensity ratings will be measured using Likert scale (0-10 rating scale, 0=not intense at all, 10=highest intensity imaginable)
Psychological Effects | Baseline to 4 weeks after drug delivery
  - Peak psychological effects will be measured by the Altered States of Consciousness (5D-ASC) questionnaire at the end of each dosing session
Psychological Effects | Baseline to 4 weeks after drug delivery
  - Peak psychological effects will be measured by the Challenging Experiences Questionnaire at the end of each dosing session
Psychological Effects | Baseline to 4 weeks after drug delivery
  - Persistent changes in attitude, mood, and behavior will be assessed using Persisting Effects Questionnaire, administered 4 weeks after each dosing session
Psychological Effects | Baseline to 4 weeks after drug delivery
  - Personality profiles will be measured using the Big Five Inventory at baseline and 4 weeks after each dosing session
Adverse Effects | Baseline to 24 hours after dosing session
  * Acute hypertension, hypotension, tachycardia, or bradycardia will be detected through blood pressure and heart rate monitoring at 10 minutes prior to drug administration and measured frequently up to 360 minutes following administration
  * Other dosing-related side effects including descriptive reports of nausea, headaches, dizziness, weakness, drowsiness, paresthesia, or blurred vision will be assessed during check-ins, after dosing effects have waned, and 24 hours following dosing

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Woolley, MD/PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bogenschutz MP, Johnson MW. Classic hallucinogens in the treatment of addictions. Prog Neuropsychopharmacol Biol Psychiatry. 2016 Jan 4;64:250-8. doi: 10.1016/j.pnpbp.2015.03.002. Epub 2015 Mar 14. PMID 25784600
- [Background] Benet-Martinez V, John OP. Los Cinco Grandes across cultures and ethnic groups: multitrait multimethod analyses of the Big Five in Spanish and English. J Pers Soc Psychol. 1998 Sep;75(3):729-50. doi: 10.1037//0022-3514.75.3.729. PMID 9781409
- [Background] Brown RT, Nicholas CR, Cozzi NV, Gassman MC, Cooper KM, Muller D, Thomas CD, Hetzel SJ, Henriquez KM, Ribaudo AS, Hutson PR. Pharmacokinetics of Escalating Doses of Oral Psilocybin in Healthy Adults. Clin Pharmacokinet. 2017 Dec;56(12):1543-1554. doi: 10.1007/s40262-017-0540-6. PMID 28353056
- [Background] Barrett FS, Bradstreet MP, Leoutsakos JS, Johnson MW, Griffiths RR. The Challenging Experience Questionnaire: Characterization of challenging experiences with psilocybin mushrooms. J Psychopharmacol. 2016 Dec;30(12):1279-1295. doi: 10.1177/0269881116678781. Epub 2016 Nov 17. PMID 27856683
- [Background] Anderson BT, Danforth A, Daroff PR, Stauffer C, Ekman E, Agin-Liebes G, Trope A, Boden MT, Dilley PJ, Mitchell J, Woolley J. Psilocybin-assisted group therapy for demoralized older long-term AIDS survivor men: An open-label safety and feasibility pilot study. EClinicalMedicine. 2020 Sep 24;27:100538. doi: 10.1016/j.eclinm.2020.100538. eCollection 2020 Oct. PMID 33150319